CLINICAL TRIAL: NCT04575480
Title: The Ideal Time Interval Between Repeated Shock Wave Lithotripsy Sessions For Renal Stones: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fadala, Fellow of urology , Urology and nephrology center , Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Urology and nephrology center
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Ideal Time Interval

STUDY DESIGN:
Intervention Model Description: Randomized trial, conducted in Urology and Nephrology Centre in Mansoura, Egypt.
  Including adults >18 years with primary single renal stone amenable for SWL according to EUA guidelines (≤ 2 cm single calyceal renal stone in a normal functioning kidney) .
  Exclusion criteria include contraindications to ESWL (uncontrolled Hypertension , coagulopathy etc), previous intervention for renal stones , congenital renal anomalies and solitary kidney.
  Patients will be randomized to one of three groups (50 Patient in each): Group 1 will undergo SWL with 3 days between each session , Group 2 will undergo SWL with 7 days between each session and Group 3 will undergo SWL with 14 days between each session. pre-ESWL and post-ESWL values will be compared.Participants will be invited after signing an informed consent including the potential risks and benefits of each intervention in this clinical study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1 (Active Comparator): Group 1 will undergo SWL with 3 days between each session.
  Interventions: Procedure: Shock Wave Lithotripsy for renal stone.
- Group 2 (Active Comparator): Group 2 will undergo SWL with 7 days between each session
  Interventions: Procedure: Shock Wave Lithotripsy for renal stone.
- Group 3 (Active Comparator): Group 3 will undergo SWL with 14 days between each session.
  Interventions: Procedure: Shock Wave Lithotripsy for renal stone.

INTERVENTIONS:
Procedure: Shock Wave Lithotripsy for renal stone. — The following protocol will be applied for all patients in study groups. SWL will be performed using the Dornier Gemini lithotripter (Dornier MedTech, Wessling, Germany) . A total of 3 000 shocks will be delivered at 80 shocks/min. The patient will receive 1 mg/kg pethidine i.v. for analgesia. Treatment will begin at machine power step 1, which will deliver 49 MPa focal pressure and 0.35 mJ/mm2. Power will be gradually increased by one step for each 200 shocks up to step 4, which deliver 70 MPa and 0.7 mJ/mm2. The maximum session number will be 3 session. Patient treated with <2 sessions will be excluded from the analysis

SUMMARY:
There is no consensus about the required time intervals between repeated SWL sessions applied for renal stones with some centers waiting for 3 days, others for one week and others up to one month to repeat lithotripsy. In the 2019 EUA guidelines stated that "There are no conclusive data on the intervals required between repeated SWL sessions. However, clinical experience indicates that repeat sessions are feasible (within 1 day for ureteral stones).

The intense use of ESWL currently, the lack of knowledge about acute lesions caused by re-treatment within a short time interval and the empirical way by which treatment is conducted, stimulated us to search for a precise answers to the question What the ideal time interval between SWL sessions in the treatment of renal stone patients should be.

This randomized controlled trial will be conducted at Urology and Nephrology Center in Mansoura, Egypt. Patients more than 18 years old with single primary renal stone fulfilling inclusion criteria will be randomly allocated to 3 groups (50 patients each).Group 1 will undergo SWL with 3 days between each session. Group 2 will undergo SWL with 7 days between each session and Group 3 will undergo SWL with 14 days between each session.

Study parameters will be renal damage including the following items:

* Tubular damage will be assessed through estimation of changes in urinary excretion of renal tubular enzyme kidney injury molecule 1(KIM-1).
* Glomerular damage will be assessed by estimation of proteinuria and changes in GFR calculated by renal isotope scan.
* Renal morphological and haemodynamic changes.
* Treatment success is defined as clinically insignificant residual fragments less than 4 mm size.

DETAILED DESCRIPTION:
STUDY DESIGN:

Randomized Trial

STUDY SETTING/LOCATION:

The study will be conducted in a single tertiary center, Urology and Nephrology Centre in Mansoura, Egypt.

STUDY POPULATION:

Adults (>18years) with primary single renal stone amenable for SWL according to EUA guidelines (C. TÜRK, 2019) .

Inclusion criteria Adult patient with ≤ 2 cm single calyceal renal stone in a normal functioning kidney.

Exclusion criteria:

1. Contraindications to ESWL:

   * Uncontrolled Hypertension
   * Renal insufficiency
   * Diabetic patient
   * Coagulopathy
   * Morbid obesity
   * Upper urinary tract obstruction
   * Active urinary tract infection
2. Previous surgical or SWL treatment of renal stones.
3. Congenital renal anomalies and solitary kidney
4. Pediatric patients (age <18 years). STUDY GROUPS Patient fulfilling the study criteria will be randomly allocated to one of three groups (50 Patient in each): Group 1 will undergo SWL with 3 days between each session. Group 2 will undergo SWL with 7 days between each session and Group 3 will undergo SWL with 14 days between each session.

Each patient will serve as internal control through comparing both pre-ESWL and post-ESWL values of our study parameters. / Candidates Potential participants will be invited to participate in this study after signing an informed consent. Potential participants will be given enough information, in a way they will understand, about the potential risks and benefits of being involved in this clinical study.

Baseline evaluation (Before ESWL) (S0):

Complete history and physical examination. Laboratory Investigations

Blood Samples:

Blood sample will be withdrawn Pre-ESWL (B.S0) for:

* CBC
* Serum creatinine
* Prothrombin concentration

Urine Samples:

* Samples of urine will be obtained before ESWL session(U.S0) for Urine analysis &estimation of KIM-1
* Urine culture will be obtained in cases of pyuria

Radiological investigation:

* NCCT will be performed. Stone criteria will be identified as regard to volumes, site, location, stone density and associated hydronephrosis.
* I.V.P (intravenous pyelography) will be performed if needed to exclude the presence of narrow neck calyx or stones in closed calyces.
* Dynamic renal scintigraphic scanning using technetium-99m Diethylene Triamine Pentaacetic Acid (TC-99m DTPA). The renal uptake, percentage of uptake from the injected dose, split function, ERPF, corrected glomerular filtration rate (GFR), time to peak clearance (T max), and half-time clearance will be calculated, because these parameters are helpful indicators in the evaluation of renal function.
* Functional MRI assessment to evaluate the renal tissue oxygenation using Blood-Oxygen Level Dependent (BOLD) and possible anatomical changes

Randomization Randomization will be performed using computer generated, sequentially numbered method.

Procedure technique:

The following protocol will be applied for all patients in study groups. SWL will be performed using the Dornier Gemini lithotripter (Dornier MedTech, Wessling, Germany) . A total of 3 000 shocks will be delivered at 80 shocks/min. The patient will receive 1 mg/kg pethidine i.v. for analgesia. Treatment will begin at machine power step 1, which will deliver 49 MPa focal pressure and 0.35 mJ/mm2. Power will be gradually increased by one step for each 200 shocks up to step 4, which deliver 70 MPa and 0.7 mJ/mm2. The maximum session number will be 3 session. Patient treated with <2 sessions will be excluded from the analysis.

After 1st ESWL session:

* Urine sample will be obtained 2to 4 hours after the end of the first session (U.S1) for estimation of urinary proteinuria and estimation of KIM-1
* Visual analogue scale will be compared between the study groups
* Non contrast spiral CT (low dose) will be performed before 2nd session to detect residual fragments, presence of obstruction and the need for re-treatment.
* Functional MRI assessment to evaluate the renal tissue oxygenation.

After 2nd ESWL session:

* Urine sample will be obtained after 2 to 4 hours after the second session (U.S2) for proteinuria and estimation of KIM-1.
* Visual analogue scale.
* Non contrast spiral CT (low dose will be performed before 3rd session to detect residual fragments, presence of obstruction and the need for re-treatment.
* Functional MRI assessment to evaluate the renal tissue oxygenation.

After 3 months of the treatment :

* Samples of urine will be obtained after 3 month from the start of treatment U.S3 for Urine analysis & estimation of urinary proteinuria and estimation of KIM-1
* Blood sample will be withdrawn (B.S3) for:

  * CBC
  * Serum creatinine and calculation of eGFR values
* NCCT will be done after 3 months of the last session of ESWL for detection of the stone free rate.
* Dynamic renal scintigraphic scanning using TC-99m DTPA as described before.
* Functional MRI assessment to evaluate the renal tissue oxygenation Statistical analysis Analysis of data will be performed with Statistical Package for Social Science (SPSS) software. Continuous data will be presented as mean ± SD when normally distributed and as medium and range when non-normally distributed. Categorical data will be presented as frequency and percentage. Comparison between mean ± SD between the three groups will be carried out by ANOVA test. Comparison between the median and range between the 3 groups will be performed by Kruskal -Wallis test. Comparison between categorical variables between groups will be performed using Chi-square or Fisher Exact test as appropriate. Regression analysis to estimate the best model which can predict the related kidney injury. In all comparison, a P.value < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion criteria Adult patient with ≤ 2 cm single calyceal renal stone in a normal functioning kidney.

Exclusion criteria:

1. Contraindications to ESWL:

   * Uncontrolled Hypertension
   * Renal insufficiency
   * Diabetic patient
   * Coagulopathy
   * Morbid obesity
   * Upper urinary tract obstruction
   * Active urinary tract infection
2. Previous surgical or SWL treatment of renal stones.
3. Congenital renal anomalies and solitary kidney
4. Pediatric patients (age <18 years).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
to identify the ideal time interval between SWL sessions used for treatment of renal stones and subsequent renal damage. | 3 months
  Renal damage:
  1. Tubular damage:
     Tubular damage will be assessed through estimation of changes in urinary execration of the renal tubular enzyme, Kidney injury molecule -1 (KIM-1).
  2. Glomerular damage:
     Glomerular damage will be assessed by the presence of proteinuria and changes of GFR calculated by renal isotope scan.
  3. Renal morphological and hemodynamic changes:
     * Changes will be assessed by estimation of ERPF by renal isotope scan.
     * The presence of peri-renal or subcapsular hematomas on non-contrast spiral CT.
     * Assessment of renal tissue oxygenation using functional MRI.

SECONDARY OUTCOMES:
3 months stone free rate | 3 months
  Treatment success is defined as clinically insignificant residual fragments of < 4 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
in partial fulfillment of MD Degree in urology
Supporting Information: Study Protocol
Time Frame: 2 years

REFERENCES:
- [Derived] Fadallah M, Abdelhalim A, Hashem A, Mortada WI, Ibrahim HAM, Sheir KZ, Harraz AM, El-Kenawy MR, El-Nahas AR. The Ideal Interval Between Repeated Shockwaves Lithotripsy Sessions for Renal Stones: A Randomized Controlled Trial. J Endourol. 2023 Dec;37(12):1305-1313. doi: 10.1089/end.2023.0345. PMID 37767632